CLINICAL TRIAL: NCT01555099
Title: A Phase-II, Double-blind, Placebo-controlled, Randomised, Parallel-group,Multi-centre Study to Assess the Efficacy and Safety of Two Staggered Dose Levels of Inhaled Once Daily AZD5423 or Twice Daily Budesonide for 12 Weeks in COPD Patients on a Background Therapy of Formoterol.
Brief Title: Multi-centre Study to Assess the Efficacy and Safety of AZD5423 in COPD Patients on a Background Therapy of Formoterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2340C00011; 2011-005389-39
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, FEV1, AZD5423
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AZD5423 (Experimental): New study drug
  Interventions: Drug: AZD5423
- Budesonide (Active Comparator): Comparator to which the new study drug will be compared
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): No drug to which both other arms will be compared
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5423 — oral inhaled
  Arms: AZD5423
Drug: Budesonide — oral inhaled
  Arms: Budesonide
Drug: Placebo — oral inhaled
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy and safety of two staggered dose levels of inhaled once daily AZD5423 or twice daily budesonide for 12 weeks in COPD patients on a background therapy of formoterol.

DETAILED DESCRIPTION:
A phase-II, double-blind, placebo-controlled, randomised, parallel-group,multi-centre study to assess the efficacy and safety of two staggered dose levels of inhaled once daily AZD5423 or twice daily budesonide for 12 weeks in COPD patients on a background therapy of formoterol.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to conducting any study specific procedures
* Men or women aged ≥ 40 years
* Men or post-menopausal or surgically sterile women. Women will be considered post-menopausal if they have been amenorrheic for at least 12 months, and have a follicle stimulating hormone (FSH) plasma concentration within the postmenopausal range as defined by the laboratory. Male patients should be willing to use barrier contraception, i.e. condom (with spermicide) from the day of dosing until at least 5 weeks after the last dose with the study drug.
* Clinical diagnosis of COPD for more than 1 year at Visit 1, according to GOLD guidelines
* Current maintenance therapy with LABA and/or LAMA, ICS/LABA or ICS plus LAMA combination
* Current or ex-smokers with a smoking history equivalent to at least 10 pack years (1 pack year = 20 cigarettes smoked per day for one year)
* Post-bronchodilator FEV1 ≥40 and ≤ 80% of the predicted normal value
* Post-bronchodilator FEV1/FVC <0,7
* Reversibility of airway obstruction according to reversibility test performed at visit 2, defined as an increase in FEV1 of ≥10% relative baseline after inhalation of in total 400 μg salbutamol or 1 mg terbutaline sulphate
* Chest radiography (not older than 12 months at Visit 2) not showing any pathological changes that would make the patient unsuitable for inclusion as judged by the Investigator
* Able to read and write and use the electronic devices (eDiary and electronic spirometry)
* Ability to complete an eDiary correctly. Baseline diary data had to be recorded for at least 8 (any 8) of the last 10 days of the run-in period to accept patients for randomized treatment (Randomisation Criteria at Visit 3).
* Provision of informed consent for genetic sampling and analyses. If a patient declines to participate in the pharmacogenetic research, there will be no consequence or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in the Clinical Study Protocol (CSP), as long as they consent (Inclusion criteria for patients taking part in the pharmacogenetic research)

Exclusion Criteria:

* Significant disease or disorder (eg, cardiovascular, pulmonary other than COPD, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study
* Any clinically relevant abnormal findings in clinical chemistry, haematology, urinalysis, physical examination, pulse, blood pressure or ECG at Visit 2, which, in the opinion of the investigator, may put the patient at risk because of his/her participation in the study
* Requirement for long term oxygen therapy
* An exacerbation of COPD, defined as use of oral or parenteral glucocorticosteroids or oral/parenteral antibiotics or hospitalisation related to COPD within 6 weeks of Visit 2
* Participation in or scheduled for an intensive COPD rehabilitation program
* Known or suspected hypersensitivity to study therapy or excipients of the study drug
* History of current alcohol or drug abuse or any condition associated with poor compliance as judged by the investigator
* Plasma donation within one month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening.
* Participation in any clinical study with an investigational drug or new formulation of a marketed drug in the 3 months prior to Visit 2
* Planned in-patient surgery or hospitalisation during the study
* Previous randomisation of treatment into the present study
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site)
* Previous allogeneic bone marrow transplant (Exclusion criteria for patients taking part in the pharmacogenetic research)
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection (Exclusion criteria for patients taking part in the pharmacogenetic research)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to mean of weeks 8 to 12 in pre-dose forced expiratory volume in 1 sec (FEV1) | Baseline (week 0), and at week 8, 10, and 12

SECONDARY OUTCOMES:
Percent change from baseline in twenty-four hour plasma cortisol | Baseline (week 0), and at week 4 and 12
Time to first exacerbation (hospitalisation, oral/parenteral corticosteroid, oral/parenteral antibiotics) | Baseline(week 0) and week 2, 4, 8, 10, 12 and daily by eDairy
The percent change from baseline in pre-dose hsCRP at week 4 and 12 | Baseline(week 0), and at week 4 and 12
Profile of pharmacokinetics (PK) of AZD5423 in terms of Cmax, tmax, AUC(0-24h), CL/F, Cav in subset of patients | Week 4 and 12
Number of St George's Respiratory Questionnaire (SGRQ-C) responders and Overall Score | Baseline(week 0), and at week 4 and 12
Assessment of Baseline/Transitional Dyspnea Index (BDI/TDI) Score | Baseline(week 0), and at week 4 and 12
Assessment of Breathlessness, Cough and Sputum Scale (BCSS) Score | Daily by eDairy
Absolute change from baseline to mean of week 2 and 4 pre-dose forced expiratory volume in 1 sec (FEV1) | Baseline (week 0), and at week 2 and 4.
Absolute change from baseline in pre-dose FEV1 | Baseline (week 0) and at week 2, 4, 8, 10 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Professor, Principal Investigator — Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego w Łodzi, ul. Kopcińskiego 22, 90-153, Łódź, Poland
Locations (44):
- Bulgaria (4):
  - Research Site, Doganovo
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- France (5):
  - Research Site, Brest
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Pessac
- Hungary (4):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Százhalombatta
- Italy (5):
  - Research Site, Foggia, FG
  - Research Site, Padua, PD
  - Research Site, Verona, VR
  - Research Site, Napoli
  - Research Site, Pisa
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gorzow Wlkp
  - Research Site, Lodz
  - Research Site, Proszowice
  - Research Site, Tarnów
- Russia (8):
  - Research Site, Barnaul, Russia
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Vladikavkaz
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (6):
  - Research Site, Vráble, Slovakia
  - Research Site, Bratislava
  - Research Site, Humenné
  - Research Site, Košice
  - Research Site, Spišská Nová Ves
  - Research Site, Zvolen
- Ukraine (7):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Zaporizhzhya